CLINICAL TRIAL: NCT05275764
Title: Comparison of the Efficacy of Intraocular Lens Optic Capture and In-the-bag Implantation Over 1 Year in Children With Congenital Cataract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: WDD-optic capture
Record Dates: First submitted 2022-02-19; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Congenital Cataract; Intraocular Lens Implantation; Optic Capture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- optic capture group: IOL optic was captured through the posterior continuous curvilinear capsulorhexis
  Interventions: Procedure: primary or secondary intraocular lens implantation surgery
- endocapsular group: IOL was placed in the bag
  Interventions: Procedure: primary or secondary intraocular lens implantation surgery

INTERVENTIONS:
Procedure: primary or secondary intraocular lens implantation surgery — primary or secondary intraocular lens implantation surgery

SUMMARY:
Approximately 30 eyes with congenital cataract who underwent primary or secondary intraocular lens implantation surgery at Zhejiang Eye Hospital from March 2018 to December 2020 were enrolled. According to the implantation method of IOL, patients were devided into the optic capture group and the endocapsular group. And through the clinical parameters of postoperative best corrected visual acuity (BCVA), intraocular pressure (IOP), IOL position and whether appear visual axis opacity to compare the outcome of the 2 IOL implantation methods.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 10 years diagnosed with congenital cataract
* underwent I / II IOL implantation in our hospital
* corneal diameter more than 9mm
* Good compliance

Exclusion Criteria:

* Patients with other ocular or systemic diseases
* patients whose IOL cannot be implanted in or after the capsule due to ocular conditions
* Children with a history of other ocular surgery
* Low compliance

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with congenital cataracts who underwent primary or secondary intraocular lens implantation surgery at the Eye Hospital Affiliated to Wenzhou Medical University.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
IOL position | through study completion, an average of 1 year
  The horizontal and vertical inclination of IOL
BCVA | through study completion, an average of 1 year
  best corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No